CLINICAL TRIAL: NCT05217186
Title: Associations Between Early Neonatal Neuroimaging, Hammersmith Infant Neurological Examination and General Movements Assessment in a Cohort of High Risk of Infants: One Year Follow Up
Brief Title: Associations Between Early Neonatal Neuroimaging, Hammersmith Infant Neurological Examination and General Movements
Acronym: highrisk
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU1
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Infant, Premature, Diseases; Infant Development; Neurologic Disorder; Development Delay; Infant Asphyxia; Infant, Small for Gestational Age; Infant, Newborn, Disease; Infant, Very Low Birth Weight
Keywords: Neonatal Neuroimaging; Hammersmith Infant Neurological Evaluation (HINE); General Movements (GMs); High Risk of Infants
MeSH Terms: conditions — Cerebral Palsy; Infant, Premature, Diseases; Nervous System Diseases; Learning Disabilities; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurements — All infants wirth high risk of cp will be assessed by neuroimaging and Hammersmith Neonatal Neurological Examination (HNNE) at term age, Prechtl's General movements (GMs) assessments form birth up to 3-5 months, and will be assesed by Hammersmith Infant Neurological Examination (HINE) at 2,3,6,9 and 12th months, also BAYLEY-III Infant and Toddler Development Assessment Scale (BAYLEY-III) at the 3rd, 6th, and 12th months.
  Other Names: Measurements of neurological development.

SUMMARY:
High risk infant is defined as infant with a negative history of environmental and biological factors, which can lead to neuromotor development problems. It is a heterogeneous group of premature infants born under thirty-seven weeks of age, with infants with low birth weight, term or developmental retardation for various reasons. Therefore, preterm infants with low birth weight can survive with a neurological sequelae such as cerebral palsy (CP), epilepsy, hearing and vision loss, mental retardation, speech and speech problems, and learning difficulties. The clinical diagnosis of CP, which can be observed in high-risk infants, is based on the combination of some neuroimaging and neurological examinations and assesments like neonatal imaging, general movements (GMs) and Hammersmith Infant Neurological Examination (HINE).

DETAILED DESCRIPTION:
High-risk infants may encounter many problems in terms of motor, cognitive, sensory, social, and academic development. Premature and LBW infants are at higher risk in terms of motor and cognitive development problems. Approximately 50% of these infants encounter neurodevelopmental problems. These problems are related to gestational age (GA), birth weight, brain damage occurring during the prenatal/perinatal period, and medical risk factors. Prematurity and low birth weight (LBW) are also among the most important causes of CP. Three methods with the best predictable validity that can determine CP before the adjusted age of 5-month is Magnetic Resonance Imaging (MRI), Prechtl's Assessment of General Movements (GMs), Hammersmith Infant Neurological Evaluation (HINE). In recent years, the diagnosis of high-risk of CP can be detected at 3 months with predictive validity and reliability by evaluating the quality of GMs. GMs are now considered the gold standard for early detection of CP because of its high sensitivity and specificity than MRI, cranial US and neurological evaluations. It was also found that cognitive or language skills may be inadequate in school age in patients with inadequate movement character and in the same postural patterns according to age, although GMs are normal. So new clinical care guidelines and new intervention research for infants with CP under the age of 2, needs to be shown. So this study aims to examine the associations between early neonatal neuroimaging, HINE and GMs assessment in a Cohort of High Risk of Infants with one year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Have periventricular hemorrhage, ICH stages 2, 3, 4, cystic PVL, stage 3 HIE, kernicterus, perinatal asphyxia, chronic lung disease, RDS, BPD, long-term oxygen (7 days), >24 hours mechanical ventilator (MV) support, 5th minute Apgar Score <3, neonatal sepsis, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), gestation age <32 weeks, and prematurity due to preterm/multiple births<1500 gr.

Exclusion Criteria:

* Infants with congenital malformation (Spina Bifida, Congenital Muscular Torticollis, Arthrogriposis Multiplex Congenita etc.)
* Infants diagnosed with metabolic and genetic diseases (Down Syndrome,Spinal Muscular Atrophy, Duchenne Muscular Dystrophy etc.)
* Infants still intubated and mechanical ventilator dependent at postterm 3 months.

Ages: 25 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: High risk of infants for cerebral palsy.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Neonatal Magnetic Resonance Imaging (MRI) | at term age of infants (40 weeks), one assesment
  Classification will be made according to the myelination status of the posterior internal capsule (PLIC), which is a robust marker showing the integrity of the cortical-spinal cord pathways at term.
  1. CP development is unlikely. Minor anomalies not associated with normal imaging or development of CP, such as IVH grade 1-2. PLIC is in normal view.
  2. Uncertain, SP possible but unlikely. Images show some evidence of damage, but symmetrical myelination is present in PLICs. Examples are stage 3 IVH, stroke not affecting the motor pathway, or HIE followed by lesion without basal ganglia or thalamus (BGT), hypoxic-ischemic injury without PLIC, pyramids, or perirolandic area
  3. He is very likely to develop CP. Evidence of brain damage or malformations involving abnormal motor structures/absence of myelination in PLICs. Typical examples; stage IV IVH, cystic PVL, HIE with IGT involvement, or brain malformation with motor cortex involvement and any imaging abnormal and with PLIC
Hammersmith Neonatal Neurological Examination (HNNE) | at term age of infants (40 weeks), one assesment
  HNNE Developed by Dubowitz and used for clinical and research purposes in the neurological examination of infants. The current form of the examination; Optimality scores were standardized by evaluating low-risk term and high-risk preterm infants at term age, 6-48 hours after birth. This scale consists of a standard proforma consisting of 34 items. Items in the proforma are scored between 1-3. Half points can be given to an item. High scores indicate good neurological status. This proforma; It is divided into 6 categories: tone (10), tone patterns (5), reflexes (6), movements (3), abnormal signs (3), and behavior (7).
Hammersmith Infant Neurological Examination (HINE) | Change from the baseline of the HINE score at 2, 3, 6, 9,12th month of infants
  The HINE is a simple, standardized, and scorable test for the clinical neurological evaluation of 2-to-24-month-old infants. It has 3 sections: (1) neurological examination (26 items, scored) evaluating cranial nerve function, posture, movements, tone, reflexes, and reactions, (2) motor milestones (8 items, unscored), and (3) behaviour (3 items, unscored). Each of the 26 items is scored first separately (as 0, 1, 2, or 3, half scores) and then the total score is calculated with a maximum score of 78. Higher score indicates good neurological function.
The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) | Change from the baseline of the BAYLEY-III score at 3, 6,12th month of infants
  The BSID-III is a neurocognitive assessment used to evaluate infants from 0-42 months and to monitor their development with 5 domains: cognitive, language (receptive and expressive communication), motor (fine and gross motor), social-emotional, and adaptive functions (17). The first three domains will be assessed. To allow comparison of results from the 5 domains, a composite score will be calculated for each domain (mean, 100±15). A composite score below -2 standard deviation (SD) (<70) will be considered a severe delay for all domains.
General Movement Assessment (GMs)1 | Measurement at preterm age (birth to 40weeks)
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character. They will be scored as cs-pr-n-ch. N show normal movement patterns.
General Movement Assessment (GMs)2 | Measurement between the term age to 9th weeks
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character. They will be scored as cs-pr-n-ch. N show normal movement patterns.
General Movement Assessment (GMs)3 | Measurement at fidgety periods of life (between 10th weeks to 20th weeks)
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character and then till about 20 weeks a "fidgety" character. Two specific abnormal movement patterns reliably predict CP in fidgety term: F (-): the absence of the fidgety character from 8-20 post-term weeks. Fidgety movements (FMs) are classified as (a) normal (F+), (b) absent (AF), when normal FMs are never observed and (c) abnormal (F-).

SECONDARY OUTCOMES:
demographic information1 | first day of birth
  birth age in weeks
demographic information2 | first day of birth
  birth weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Hatice Adiguzel, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No